CLINICAL TRIAL: NCT00264966
Title: A Double-blind, Placebo-controled, Crossover Study To Evaluate the Efficacy, Safety and Tolerability of Inhaled ASM8-003 in Subjects With Mild Allergic Asthma.
Brief Title: Multiple Dose ASM8 in Mild Asthmatics
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Syntara (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ASM8-003
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Asthma
Keywords: Mild asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ASM8

SUMMARY:
To determine the safety and efficacy of multiple doses of ASM8 antisense oligonucleotides in asthmatics.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, crossover trial to evaluate the safety, tolerability and efficacy of inhaled ASM8 for the treatment of allergen-induced asthma. Individuals with stable, mild to moderate allergic asthma by American Thoracic Society (ATS) criteria (1), with a history of episodic wheeze and shortness of breath, will be eligible for enrolment. The study is divided into 2 parts.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Men and women 18 to 65 years of age; generally good health; mild to moderate, stable, allergic asthma as defined by ATS criteria (1); history of episodic wheeze and shortness of breath; forced expiratory volume in 1 second (FEV1) at baseline ≥70% of the predicted value; able to comprehend and follow all required study procedures; willing and able to sign an informed consent form.

Part 2: Methacholine challenge at baseline (PC20 ≤16 mg/mL); positive skin-prick test to common aeroallergens (cat, dust mite, grass, pollen) and positive allergen-induced early and late airway bronchoconstriction.

Exclusion Criteria:

* Part 1 and Part 2: Significant acute or chronic medical or psychiatric illness; known coagulopathy, worsening of asthma or respiratory infection in the preceding 6 weeks; use of inhaled or oral corticosteroids within the last 28 days, antihistamines, immunosuppressives, nonsteroidal anti-inflammatory drugs, or anticoagulants (intermittent doses of short-acting β2-agonist are allowed); use of medications that may interact with ASM8; investigational drug use within 30 days; any clinically significant abnormality on screening laboratory determinations; current tobacco use in previous 3 months or 10 pack-years; pregnant or lactating women; women actively seeking pregnancy or who are not using adequate contraception; history of serious adverse effect (SAE) or hypersensitivity to any drug; 20% decrease in FEV1 or FVC with baseline saline in methacholine challenge during screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2005-12; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Comparison of the allergen-induced late asthmatic response (LAR) between ASM8 and placebo

SECONDARY OUTCOMES:
Evaluation of the safety and tolerability of ASM8.
Comparison of the allergen-induced early asthmatic response (EAR) between ASM8 and placebo.
Comparison of the allergen-induced airway hyperresponsiveness between ASM8 and placebo.
Comparison of the allergen-induced changes in sputum eosinophils at 7 and 24 hours post allergen, between the ASM8 and placebo.
Determination of the plasma and sputum pharmacokinetic profile of single- and repeated-doses of ASM8 in patients with mild asthma.
Determination of the pharmacodynamic activity of ASM8 on specific gene expression, protein levels, differential cell counts, and eosinophilic cationic protein (ECP), as measured in sputum samples.
Relief medication use in the ASM8 versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Paul O'Byrne, MD, Principal Investigator — McMaster University
Locations (3):
- Canada (3):
  - McMaster University, Hamilton, Ontario
  - Hopital Laval, Ste-Foy, Quebec
  - Saskatoon Hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Gauvreau GM, Boulet LP, Cockcroft DW, Baatjes A, Cote J, Deschesnes F, Davis B, Strinich T, Howie K, Duong M, Watson RM, Renzi PM, O'Byrne PM. Antisense therapy against CCR3 and the common beta chain attenuates allergen-induced eosinophilic responses. Am J Respir Crit Care Med. 2008 May 1;177(9):952-8. doi: 10.1164/rccm.200708-1251OC. Epub 2008 Jan 31. PMID 18244953